CLINICAL TRIAL: NCT05810831
Title: Efficacy of Massage Versus Massage With Post Isometric Relaxation Exercises in Temporomandibular Disorder
Brief Title: Efficacy of Massage Versus Massage With Post Isometric Relaxation Exercises in Temporomandibular Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/521
Record Dates: First submitted 2023-03-15; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Pain, Joint
MeSH Terms: conditions — Arthralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage with post isometric relaxation exercises (Experimental)
  Interventions: Diagnostic Test: Massage with post isometric relaxation exercises
- Massage (Experimental)
  Interventions: Diagnostic Test: Massage

INTERVENTIONS:
Diagnostic Test: Massage with post isometric relaxation exercises — Post isometric relaxation will be performed in supine position with neutrally positioned head.
  Arms: Massage with post isometric relaxation exercises
Diagnostic Test: Massage — conservative physiotherapy protocol including massage
  Arms: Massage

SUMMARY:
To determine effectiveness of massage versus massage with post isometric relaxation exercises in temporomandibular disorders for pain and limited joint mobility.

ELIGIBILITY:
Inclusion Criteria:

* patients with clinical features with myofascial pain and limited mouth opening fulfilling the Axis Group I of RDC/TMD criteria,
* absence of temporomandibular disc displacement with or without reduction,
* good general health (absence of chronic diseases which may affect temporomandibular joint or the masticatory muscles),
* full dental arches with natural teeth or missing teeth replaced with fixed dental prostheses

Exclusion Criteria:

* earlier splint therapy,
* pharmacotherapy (e.g., hormone replacement therapy, oral contraception and antidepressants),
* injury of masticatory organ,
* undergoing orthodontic treatment,
* inflammation in oral cavity (e.g., impacted molars and pulp inflammation) and fibromyalgia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Massage exercises , Massage with post isometric relaxation exercises | 6 Months

IPD SHARING:
Plan to Share IPD: No